CLINICAL TRIAL: NCT03624582
Title: Validity and Reliability of the Activity Preference Assessment: A Shape Up Kids Ancillary
Brief Title: Shape Up Kids Fitness Ancillary
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Louisiana State University, Baton Rouge (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, S. Nicole Fearnbach, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: 2018-028; P30DK072476 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-08-10 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Childhood Obesity
Keywords: Cardiorespiratory fitness; Sedentary behavior; Physical activity; Decision-making; Cardiometabolic risk factors
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of this study is to quantify the decision-making process and underlying biases around leisure activity behaviors using the Activity Preference Assessment (APA), a novel psychological task. The investigators plan to validate the APA against objectively measured sedentary and physical activity time, and examine its potential to predict health-related outcomes in children and adolescents. The Shape Up Kids Fitness Ancillary protocol will add exercise testing, cognitive and behavioral measures, accelerometry, and questionnaires to the existing Shape Up Kids primary study dataset.

DETAILED DESCRIPTION:
The investigators will enroll 60 boys and girls (50% female) between the ages of 8-17 years into this pilot and feasibility ancillary study. The aims of this study are to validate and test the reliability of the Activity Preference Assessment (APA), as described below.

Aim 1: To examine the convergent validity of the APA against habitual physical and sedentary activity time measured objectively by seven days of accelerometry, as well as leisure activity choices during a 30-minute free-choice play period.

Aim 2: To examine the criterion validity of the APA against concurrent measures of body composition, cardiometabolic health indicators, aerobic fitness, and physical strength.

Aim 3: To measure the test-retest reliability of APA outcomes through repeated measures separated by approximately one week.

Exploratory Aim: To investigate patterns or clusters of activity preferences through exploratory factor analysis of activity liking VAS scores.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the Shape Up Kids primary study
* Height ≥ 4 feet 8 inches
* Body weight < 350 lbs

Exclusion Criteria:

* American College of Sports Medicine (ACSM) contraindications to exercise testing (i.e., medical history of cardiovascular or pulmonary conditions, physical conditions that affect the ability to exercise)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will identify and recruit 60 participants from the Shape Up Kids primary study sample of 360 participants. Ancillary participants will be between the ages of 8-17 years. We will have an even distribution of boys (n=30) and girls (n=30) and aim to have a representative distribution of race.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Time 1 APA bias scores | Day 0 / Primary Study Visit
  Bias scores are calculated from reaction times and choices made during the forced-choice section of the APA. Scores range from -100 to +100, with negative scores indicating a bias towards physical activities, and positive scores indicating a bias towards sedentary activities.
Time 2 APA bias scores | 8-21 days after Primary Study Visit
  Bias scores are calculated from reaction times and choices made during the forced-choice section of the APA. Scores range from -100 to +100, with negative scores indicating a bias towards physical activities, and positive scores indicating a bias towards sedentary activities.
Habitual physical and sedentary activity | 7 days between visits
  Physical and sedentary activity time are measured for 24 hours per day over 7 consecutive days, including 2 weekend days, using ActiGraph GT3X+ accelerometers worn on the left mid-axillary line.
Free-choice play period | 8-21 days after Primary Study Visit
  Children will have 30 minutes to play freely in a room with a variety of sedentary and physical activity choices. Trained observers will record children's activity every 15 seconds.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 8-21 days after Primary Study Visit
  Cardiorespiratory fitness, or VO2peak in mL/kg/min, is measured using a graded cycle ergometer test to volitional fatigue.
Body composition 1 | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, body composition is measured using bioelectrical impedance analysis (BIA).
Body composition 2 | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, body composition is measured using whole-body dual-energy x-ray absorptiometry (DXA).
Body composition 3 | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, body composition is measured using whole-body magnetic resonance imaging (MRI).
Physical strength | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, physical strength is assessed with dynamometers.
Resting blood pressure | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, blood pressure is assessed after 5 minutes of rest.
Resting heart rate | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, heart rate is assessed after 5 minutes of rest.
Cardiometabolic disease biomarkers | Day 0 / Primary Study Visit
  In the Shape Up Kids primary study, fasting levels of lipid, glucose, and inflammatory biomarkers are assessed via blood draw with a single Chem 26 assay panel.
Time 1 activity liking and wanting Visual Analog Scale (VAS) scores | Day 0 / Primary Study Visit
  Participants will rate how much they like to do and want to do each of the activities included in the APA on VAS that range from 0 or "Not at all" to 100 or "Like/Want very much"
Time 2 activity liking and wanting VAS scores | 8-21 days after Primary Study Visit
  Participants will rate how much they like to do and want to do each of the activities included in the APA on VAS that range from 0 or "Not at all" to 100 or "Like/Want very much"

OTHER OUTCOMES:
International Sedentary Assessment Tool | 8-21 days after Primary Study Visit
  Children will fill out questionnaires regarding possible socio-emotional factors that can influence activity choices, including the International Sedentary Assessment Tool. This survey will be scored according to standard published procedures.
Mood and Feelings Questionnaire | 8-21 days after Primary Study Visit
  Children will fill out questionnaires regarding possible socio-emotional factors that can influence activity choices, including the Mood and Feelings Questionnaire (short version). This survey will be scored according to standard published procedures.
Physical Self Description Scale | 8-21 days after Primary Study Visit
  Children will fill out questionnaires regarding possible socio-emotional factors that can influence activity choices, including the Physical Self Description Scale. This survey will be scored according to standard published procedures.
Body Esteem Scale | 8-21 days after Primary Study Visit
  Children will fill out questionnaires regarding possible socio-emotional factors that can influence activity choices, including the Body Esteem Scale. This survey will be scored according to standard published procedures.
Neighborhood and home environment survey | 8-21 days after Primary Study Visit
  Parents will describe environmental factors through a neighborhood and home environment survey. Selected items from this survey will be used as covariates in analyses.

CONTACTS AND LOCATIONS:
Overall Officials: S. Nicole Fearnbach, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearnbach SN, Martin CK, Heymsfield SB, Staiano AE, Newton RL Jr, Garn AC, Johannsen NM, Hsia DS, Carmichael OT, Ramakrishnapillai S, Murray KB, Blundell JE, Finlayson G. Validation of the Activity Preference Assessment: a tool for quantifying children's implicit preferences for sedentary and physical activities. Int J Behav Nutr Phys Act. 2020 Aug 24;17(1):108. doi: 10.1186/s12966-020-01014-6. PMID 32831103